CLINICAL TRIAL: NCT00953199
Title: A Single Center, Randomized, Double-Blind Controlled Study of Topical Endoluminal Pancreatic Duct Lidocaine for Prevention of Post-ERCP Pancreatitis
Brief Title: Topical Pancreatic Duct Lidocaine for Prevention of Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abraham Mathew MD (Other)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor-Investigator, Abraham Mathew MD, Professor of Medicine, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Lidocaine
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Pancreatitis
Keywords: endoscopic retrograde cholangiopancreatography; ERCP; pancreatitis; lidocaine; post-ERCP pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidocaine (Experimental): Study subjects receive a 1:1 combination of 5 ml Diatrizoate 60% and 5 ml Lidocaine Hydrochloride 2%
  Interventions: Drug: Lidocaine Hydrochloride
- Normal Saline (Active Comparator): The control arm receives a 1:1 combination of 5 ml Diatrizoate and 5ml saline.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — 1:1 combination of contrast dye Diatrizoate 60% (5 ml) diluted with lidocaine 2% (5 ml) used at ERCP. Lidocaine will only be used once, and thus a maximum dose of 100 mg will be employed. If the patient requires more contrast agent, this will be used without the addition of lidocaine.
  Arms: Lidocaine
Drug: Normal Saline — 1:1 combination of contrast dye Diatrizoate 60% (5 ml) diluted with normal saline 0.9% (5 ml) used at ERCP (standard of care).
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to determine if lidocaine is effective in reducing the incidence of post-ERCP pancreatitis.

DETAILED DESCRIPTION:
Post endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis is a common cause of morbidity for which there is no known pharmacologic prophylaxis. Post-ERCP pancreatitis is thought to be caused by several factors, including intraductal pressure, multiple duct injections with contrast, and neural arc reflexes. Lidocaine is a safe, inexpensive class IV antiarrhythmic that has topical anesthetic effects, inhibits trypsin activity, and may potentially prevent post-ERCP pancreatitis by injection directly into the pancreatic duct at the time of ERCP. Lidocaine has been shown to inhibit phospholipase A2, a key pancreatic enzyme, interrupt local arc reflexes to stop neuronal transmission, and to dampen GI tract mucosal reflexes to prevent high ductal pressure.

The key objective of this study is to determine if injection of lidocaine is beneficial in preventing post-ERCP pancreatitis. Subjects will be randomized to study group or control group in an equal ratio. The physicians performing the ERCP will be unaware of the treatment group to which patients have been assigned. Study arm will receive contrast agent Diatrizoate 60% (5 ml) diluted with lidocaine 2% (5 ml) during ERCP. Control arm will receive contrast agent Diatrizoate 60% (5 ml) diluted with normal saline 0.9% (5 ml) during ERCP. Diatrizoate diluted with normal saline is the standard of care. Patients will be contacted 1 day and 1 week post-ERCP to assess for symptoms of pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients included are >18 years old, referred to Endoscopy Clinic for an ERCP for any well established indication such as: biliary strictures, benign and malignant hepato-pancreato-biliary tumors, chronic pancreatitis, and suspected sphincter of Oddi dysfunction

Exclusion Criteria:

* Known sensitivity to lidocaine or contrast agent
* History of seizure disorder
* History of cardiac arrhythmia (tachyarrhythmia, bradyarrhythmia, cardiac conduction defects, prolonged QT syndrome)
* History of congestive heart failure
* Active acute pancreatitis before procedure
* Planned biliary stent removal without pancreatogram
* Pregnancy
* Incarcerated individuals
* Less than 18 years of age
* Previous sphincterotomy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Mathew, M.D., M.S., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosen-Binker LI, Binker MG, Negri G, Tiscornia O. Acute pancreatitis possible initial triggering mechanism and prophylaxis. Pancreatology. 2003;3(6):445-56. doi: 10.1159/000074972. Epub 2003 Nov 19. PMID 14631103
- [Background] Kiyonari Y, Nishina K, Mikawa K, Maekawa N, Obara H. Lidocaine attenuates acute lung injury induced by a combination of phospholipase A2 and trypsin. Crit Care Med. 2000 Feb;28(2):484-9. doi: 10.1097/00003246-200002000-00033. PMID 10708188
- [Background] Makela A, Kuusi T, Schroder T. Inhibition of serum phospholipase-A2 in acute pancreatitis by pharmacological agents in vitro. Scand J Clin Lab Invest. 1997 Aug;57(5):401-7. doi: 10.3109/00365519709084587. PMID 9279965
- [Background] Portiansky EL, Gonzalez PH. Protective effect of lidocaine in the experimental foot-and-mouth disease pancreatitis. Experientia. 1995 Nov 15;51(11):1060-2. doi: 10.1007/BF01946916. PMID 7498445
- [Background] Schroder T, Kinnunen PK, Lempinen M. Xylocaine treatment in experimental pancreatitis in pigs. Scand J Gastroenterol. 1978;13(7):863-5. doi: 10.3109/00365527809182204. PMID 725507
- [Background] Schwartz JJ, Lew RJ, Ahmad NA, Shah JN, Ginsberg GG, Kochman ML, Brensinger CM, Long WB. The effect of lidocaine sprayed on the major duodenal papilla on the frequency of post-ERCP pancreatitis. Gastrointest Endosc. 2004 Feb;59(2):179-84. doi: 10.1016/s0016-5107(03)02540-9. PMID 14745389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2010 -May 2013, recruited from the endoscopy unit
Period: Overall Study
Arm/Group | Lidocaine | Normal Saline
Started | 254 | 252
Completed | 254 | 252
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult patients send for ERCP with a chance of contrast injection into the pancreatic duct
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Normal Saline | Total
Number analyzed (Participants) | 254 | 252 | 506
Age, Continuous [Mean (Full Range); unit: years] | 56 [18 to 99] | 55.6 [19 to 92] | 55.8 [18 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 126 | 254
  Male | 126 | 126 | 252

OUTCOME MEASURES:

1. Primary Outcome: Post ERCP Pancreatitis is the Primary Outcome.
Description: The primary outcome of interest will be development of acute pancreatitis defined as new or worsening abdominal pain post-ERCP associated with an increase in serum amylase at least 3 times the upper limit of normal.
Time Frame: 24-48 hours post-procedure
Measure: Number; unit: participants
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 254 | 252
participants | 26 | 20
Statistical Analysis 1: Comparison: Lidocaine vs Normal Saline; We calculated the sample size to be 570 in each arm, providing 80% power, allocation 1:1, two-sided, alpha 0.05, withdrawal rate of 3% and a reduction in pancreatitis from 8% to 4%. Randomization is performed with permuted blocks of 20. Analysis is based on intention to treat; Test type: Superiority or Other; p = .45, Chi-squared — .05 was set as level of significance

2. Secondary Outcome: Serum Amylase Levels
Description: serum amylase levels are measure by a blood draw
Time Frame: measurement is taken 2 hrs after ERCP
Measure: Mean (Full Range); unit: units/liter
Arm/Group | Lidocaine | Normal Saline
Number analyzed (Participants) | 254 | 252
units/liter | 130 [30 to 1826] | 128 [30 to 4000]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 48 hrs. Patients are observed in the recovery area until they are discharged after ERCP or admitted, usually about 2-3 hrs. They are called after 24 -48 hrs and later after a week for follow up.
Description: Pancreatitis and its symptoms were the study outcomes and not considered here as a separate adverse event
Arm/Group | Lidocaine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/254 | 0/252
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/252
Other Adverse Events (participants affected / at risk) | 0/254 | 0/252

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No